CLINICAL TRIAL: NCT01579188
Title: A Double-blind, Multicenter, Randomized Phase III Study of the Telomerase Vaccine, GV1001 Administered After Curative Intent Chemo-radiotherapy in Patients With Inoperable Stage III Non-small Cell Lung Cancer Compared to Best Supportive Care
Brief Title: Study of the Telomerase Vaccine GV1001 to Treat Patients With Inoperable Stage III Non-small Cell Lung Cancer
Acronym: LucaVax
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kael-GemVax Co., Ltd. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KG 1/2012
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Inoperable Stage III Non-small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: interventions — GV1001 peptide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GV1001 (Experimental): The adjuvant GM-CSF is administered first as an intradermal injection followed in 10-15 minutes by the GV1001 peptide injected into the same site.
  Interventions: Drug: GV1001
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: GV1001 — Intradermal injection 0.84 mg ± 0.084 mg 3 times in Week 1 (Monday, Wednesday, and Friday) and once (Mondays) in Weeks 2, 3, 4, 6, 8, and 10, followed by boost injections given on Weeks 14, 18, 22, 26, and thereafter at 12 week intervals up to Week 98
  Arms: GV1001
Drug: normal saline — two injections of normal saline injected in the same manner as the experimental drug, GV1001
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate survival in inoperable stage III Non-small Cell Lung Cancer patients following chemo-radiotherapy followed by GV1001 vaccination plus best supportive care.

DETAILED DESCRIPTION:
Lung cancer (both small cell and non-small cell) is the second most common cancer in both men (after prostate cancer) and women (after breast cancer). It accounts for about 15% of all new cancers. Lung cancer is the world's leading cause of cancer death with more than 1.6 million new cases diagnosed each year.

About 85 percent of lung cancer patients have Non-small Cell Lung Cancer (NSCLC ) and are usually diagnosed with advanced disease and have few treatment options and a very low survival rate.

Radiotherapy is the treatment of choice in the successful treatment of stage III NSCLC. However, the 5-year survival for stage III patients treated with radiotherapy alone is less than 10%. Several types of chemotherapy treatments have been investigated, however, progress has been limited. Most patients die from relapsed disease.

The peptide telomerase vaccine, GV1001, is under development for use as active immunotherapy in the treatment of cancer. Normally, the immune system is tolerant to self-proteins and peptides, while being able to react to foreign pathogens. However, cancer cells are degenerated cells and many of their peptides and proteins are self-proteins or peptides. By using vaccination, the immune tolerance towards a specific peptide or protein can be circumvented.

ELIGIBILITY:
Inclusion Criteria:

Patients may be entered in the study only if they meet all of the following criteria:

1. Male or female patient ≥ 18 years of age;
2. Histologically or cytologically confirmed inoperable NSCLC stage III disease;
3. Patient must have received chemo-radiotherapy with a curative intent with the following definition: any planned regimen consisting of a platinum-doublet containing chemotherapy given concomitantly with up to 66Gy of radiation therapy. Gemcitabine cannot be part of the platinum-based doublet;
4. Life expectancy of ≥ 3 months;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2;
6. Patients must have adequate bone marrow function as evidenced by absolute neutrophil count (ANC) ≥ 1.0 X 109/L, hemoglobin ≥ 9.0 g/dL (a hemoglobin < 9.0 g/dL at Screening is acceptable if it is corrected to ≥ 9 g/dL by growth factor or transfusion prior to first dose), and platelet count ≥ 75 X 109/L (platelet counts below 75 X 109/L may be re-screened within 4 weeks of chemoradiotherapy);
7. Patients must have adequate liver function as evidenced by bilirubin ≤ 1.5 times the upper limit of the normal range (ULN), and alkaline phosphatase, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 X ULN;
8. Female patients of childbearing potential (i.e. ovulating, premenopausal, not surgically sterile), and all male patients are required to be sexually abstinent or use a medically accepted contraceptive regimen during their participation in the study and for 90 days after study completion. Medically accepted contraceptive methods are defined as those with 90% or greater efficacy;
9. Females of childbearing potential must have a negative pregnancy test;
10. Females may not be breastfeeding; and
11. Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

Patients will not be entered in the study for any of the following reasons:

1. Prior treatment with gemcitabine, prior targeted therapy (including erlotinib [Tarceva®], or gefitinib [Iressa®]), or immunological therapy including tumor vaccine therapy intended for the management of NSCLC;
2. A minimum of 1 week and a maximum of 4 weeks must have elapsed from the chemo-radiotherapy and patient must have recovered from all treatment-related toxicities to Grade ≤ 1 (CTCAE version 4.03), except for alopecia;
3. History of other malignancies except: (1) adequately treated basal or squamous cell carcinoma of the skin; (2) curatively treated, a) in situ carcinoma of the uterine cervix, b) prostate cancer, or c) superficial bladder cancer; or (3) other curatively treated solid tumor with no evidence of disease for ≥ 3 years;
4. Received treatment in another clinical study within the 30 days prior to commencing study treatment or patients who have not recovered from side effects of an investigational drug to Grade ≤ 1 (CTCAE version 4.03), except for alopecia;
5. Are currently receiving any other cancer treatment, even if given with palliative intent;
6. Uncontrolled pleural effusions, ascites, or other third space fluid collections;
7. Uncontrolled diabetes mellitus Type 1 or 2;
8. Significant cardiovascular impairment (history of congestive heart failure > New York Heart Association (NYHA) Grade II, unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia);
9. Patients with organ allografts requiring immunosuppression;
10. Need for systemic steroid treatment unless chronic daily dose used is ≤ 5mg prednisone or equivalent. Note: Higher dose systemic steroid treatment (≥ 60mg/day of prednisone or equivalent) administered for ≤ 2 weeks in any single episode is permissible if administered for an acute inflammatory condition;
11. Known severe adverse reactions to vaccines;
12. Known severe adverse events or allergy to GM-CSF;
13. Known positive human immunodeficiency virus (HIV), known hepatitis B surface antigen, or hepatitis C positive; and
14. Have any medical condition that would interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years
  To evaluate OS in inoperable stage III NSCLC patients following chemoradiotherapy administered with a curative intent followed by GV1001 vaccination plus best supportive care (BSC)

SECONDARY OUTCOMES:
Safety and tolerability of GV1001 | 2 years
  To evaluate the safety and tolerability of GV1001, progression-free survival (PFS), and QoL using the general EuroQoL Five Dimensional Questionnaire (EQ-5D) and the Lung Cancer Symptom Scale (LCSS).
Immunological response | 2 years
  To evaluate the immunological response parameters as measured by T- cell functional assays and T-cell sub-population analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Sinae Jeong, Study Director — Kael-GemVax Co., Ltd.